CLINICAL TRIAL: NCT02678936
Title: Anal fistUla Repair With Platelet-Rich plasmA (AURoRA)
Brief Title: Anal Fistula Repair With Platelet-rich Plasma
Acronym: Aurora
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aurora
Record Dates: First submitted 2014-12-19; First posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Rectal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP (Experimental): The operation will be performed with application of platelet rich plasma
  Interventions: Biological: PRP
- non-PRP (No Intervention): The operation will be performed without addition of platelet-rich plasma

INTERVENTIONS:
Biological: PRP — Application of platelet-rich plasma during surgery
  Arms: PRP

SUMMARY:
Anal fistula is a very common disease with a high impact on life quality. The only commonly accepted treatment option is surgery. A wide range of operations and techniques have been developed all suffering from a relatively high recurrence rate.

The investigators propose the combination of the mucosal advancement flap with application of platelet-rich plasma (PRP) in the fistulectomy site. This study aims to test the hypothesis that by applying PRP the healing rate of complicated anal fistulas can be improved in comparison to a control group where the operation is performed without addition of PRP.

ELIGIBILITY:
Inclusion Criteria:

* complicated anal fistula with patient fit for surgical treatment
* minimum 6 weeks after
* written informed consent

Exclusion Criteria:

* age <18
* pregnancy
* drug abuse, drug substitution program
* homeless (follow-up difficult)
* restricted in legal capacity
* simple fistulas requiring fistulotomy
* complicated fistulas requiring an anus praeter naturalis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Healing rate | 2 Years

SECONDARY OUTCOMES:
Influence of risk factor smoking on healing rate | 2 years
Influence of risk factor high BMI on healing rate | 2 years
Influence of risk factor chronic renal failure on healing rate | 2 years
Influence of sex on healing rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Lorenz, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital of Basel, Basel, Switzerland